CLINICAL TRIAL: NCT06710145
Title: The Effect of Using the Combat Attention App on the Risk of Post-traumatic Symptoms
Status: Not yet recruiting | Type: Observational
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Other Study IDs: TAU-Combat-Attention
Record Dates: First submitted 2024-10-31; First posted 2024-11-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: PTSD - Post Traumatic Stress Disorder
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Attention App Users: Soldiers who used the App and completed at least one training session
  Interventions: Behavioral: Combat Attention Training
- Non Users: Soldiers matched on age, sex, and specialty to the Attention App Users group who never used the App

INTERVENTIONS:
Behavioral: Combat Attention Training — The Combat Attention App is a response-time based mechanized preventive intervention designed to train combat soldiers' attention toward threats before combat exposure in order to reduce the risk for combat-related post-trauma symptoms. In light of the results of controlled studies that proved the efficacy of this preventive intervention, the Israel Defense Forces (IDF) decided at the beginning of the Iron Swords War (October 7th, 2023) to implement an internet-based App of the intervention, and soldiers and combat reservists were invited to train on the Combat Attention App.
  Groups: Attention App Users

SUMMARY:
Military service and reserve duty in combat units entails exposure to traumatic events that require mental adjustment. In light of the results of controlled studies that proved the effectiveness an response-time based mechanized training protocol in reducing risk for post-trauma symptoms in deployed combat soldiers, the Israeli Defense Forces decided at the beginning of the Iron Swords War to implement an internet-based App of the intervention. Soldiers and combat reservists were invited to use the Combat Attention App. The purpose of this study is to examine the effectiveness of the Combat Attention App in relation to a control group of soldiers who did not use the App in reducing risk for post-traumatic stress symptoms of deployed soldiers.

DETAILED DESCRIPTION:
Participants who used the Combat Attention App before combat deployment and a group of matched (age and sex) participants who did not use the App will be compared on PTSD, depression, and anxiety symptoms post deployment.

ELIGIBILITY:
Inclusion criteria:

* Age over 18 years.
* Served as an enlisted soldier or reservist during the Iron Swards War.
* Used the Combat Attention App or can serve as a matched control who did not use the App.
* Colloquial Hebrew sufficient to fill out the research questionnaires.

Exclusion criteria:

* Below 18 years of age.
* Colloquial Hebrew that is insufficient to fill out the research questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of enlisted and reservist soldiers who participated in the Iron Swards war and either used or did not use the attention App.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | January-June 2025
  Measures PTSD symptoms according to DSM-5
IDF Medical Records | January-June 2025
  Holds all the medical information and contact with health/mental health professionals during one's service

SECONDARY OUTCOMES:
Combat Experiences Scale | January-June 2025
  Measures the occurrence of specific combat events
Patient Health Questionnaire 9 (PHQ-9) | January-June 2025
  Measures Depression symptoms according to DSM-5
Attention Bias Questionnaire (ABQ) | January-June 2025
  Measures subjective experiences of attention allocation to threats
GAD-7 | January-June 2025
  measures symptoms of generalized anxiety disorder
Dissociative Experiences Scale (DES) | January-June 2025
  measures dissociative symptoms associated with trauma exposure

CONTACTS AND LOCATIONS:
Overall Officials: Yair bAR-hAIM, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wald I, Fruchter E, Ginat K, Stolin E, Dagan D, Bliese PD, Quartana PJ, Sipos ML, Pine DS, Bar-Haim Y. Selective prevention of combat-related post-traumatic stress disorder using attention bias modification training: a randomized controlled trial. Psychol Med. 2016 Sep;46(12):2627-36. doi: 10.1017/S0033291716000945. Epub 2016 Jul 5. PMID 27377418